CLINICAL TRIAL: NCT00502268
Title: A Prospective, Randomized, Open-Label Trial Investigating the Effect of 1 Alpha Hydroxy Vitamin D2 on the Development of Coronary Calcification in New ESRD Patients Using the 1-84/7-84 PTH Ratio to Determine Dosing
Brief Title: Vitamin D and Carboxy PTH Fragments in Coronary Calcification
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study never initiated
Sponsor: Southeast Renal Research Institute (Other)
Responsible Party: Principal Investigator, James A. Tumlin MD, Nurse, Southeast Renal Research Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SBPTH-CC1
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Coronary Calcification; Endstage Renal Disease; Parathyroid Hormone
Keywords: Coronary Calcification; Endstage Renal Disease; Parathyroid hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Placebo Comparator): Doxercalciferol administration by DOQI and 2nd Gen PTH assay
  Interventions: Drug: Doxercalciferol administration
- Group 2 (Active Comparator): Doxercalciferol administered by 1-84-7-84 ratio between 1.4-1.6
  Interventions: Drug: Doxercalciferol administered by 1-84-7-84

INTERVENTIONS:
Drug: Doxercalciferol administration — Doxercalciferol administration
  Arms: Group 1
Drug: Doxercalciferol administered by 1-84-7-84 — Doxercalciferol administered by 1-84-7-84
  Arms: Group 2

SUMMARY:
Arterial calcification within the coronaries and other vessels is greatly accelerated among patients with chronic or end-stage kidney disease. The mechanisms leading to increased calcification are unknown, but include hyperphosphatemia, hyperparathyroidism and altered vitamin D metabolism. Moreover, recent data demonstrates that circulating carboxy fragments of PTH (7-84) are physiologic antagonists of intact PTH (1-84) and may directly contribute to vascular calcification. Current PTH assays no not distinguish between intact and carboxy PTH fragments leading to an overestimation of intact PTH levels. Because second generation PTH assays detect both 1-84 and 7-84 PTH fragments, the use of vitamin D analogues to treat secondary hyperparathyroidism could lead to excessive suppression of 1-84 and a preponderance of carboxy PTH fragments. Moreover, increased administration of vitamin D analogues amy contribute to vascular calcifications. To investigate these questions, we plan to investigate the effect of managing new ESRD patients using conventional and third generation PTH assays on vitamin D administration and the development of coronary calcification. Hypothesis #1: Clinical management of secondary hyperparathyroidism in new hemodialysis patients using the Scantibodies 1-84/7-84 PTH ratio for one year will reduce the amount of Vitamin D administration resulting in reduced coronary calcification compared to patients in which PTH management is accomplished by conventional, second generation PTH assay.

DETAILED DESCRIPTION:
Patients with chronic renal failure are at increased risk for vascular calcification and cardiovascular complications. For example, data from the USRDS database demonstrates that 42% of all deaths among chronic dialysis patients are cardiovascular in origin with 22% of those deaths due to arrhythmias or overt acute myocardial infarction. While numerous factors including hypertension, hyperlipidemia and diabetes contribute to both renal failure and coronary disease, recent studies find that patients with CKD experience an accelerated rate of coronary calcification. Medial calcification reduces compliance of medium to large elastic arteries such as the aorta and common carotids. The resulting loss of elasticity is thought to contribute to the high prevalence of systolic hypertension and left ventricular hypertrophy (LVH) among patients with ESRD 15.

The type of vascular calcification associated with diabetes and ESRD is histologically distinct from that found in atherosclerotic plaques. In patients with CKD or diabetes calcium deposits are concentric and uniformly distributed within the medial layer of the vessel wall. The deposition of calcium does not require the presence of atherosclerotic lesions and occurs in the absence of intimal hyperplasia. Infiltration of the adventia by T cells and activated macrophages leads to expression of bone morphogenetic protein 2 (BMP-2) and osteopontin (OPN) by pericytic myofibroblasts. In diabetics, BMP-2 expression is enhanced by the simultaneous upregulation of two BMP-2 associated transcription factors Msx1 and Msx2 3. The resulting transcription of BMP-2 genes leads to mineralization of non-endochondrial matrix. The expression of OPN is a consistent feature of medial calcification 4. Osteopontin or "bone bridge" is a highly phosphorylated glycoprotein that binds calcium and integrin receptors. The expression of osteopontin can be stimulated by vitamin D and increased circulating levels of phosphate.

Moreover, physiologic concentrations of 1, 25, dihydroxyvitamin D increases calcium deposition in cultured vascular smooth muscle cells and is associated with reduced expression of PTH related peptide (1-34 PTH) suggesting that amino PTH fragments are not only involved in regulating bone turnover, but also function to prevent dystrophic vascular calcification. Indeed, these observations raise the question of whether carboxy PTH fragments can accelerate vascular calcification.

Because second generation PTH assays detect both 1-84 and 7-84 PTH fragments, the use of vitamin D analogues to treat secondary hyperparathyroidism could lead to excessive suppression of 1-84 and a preponderance of carboxy PTH fragments. As observed by Jono et.al accumulation of 7-84 could contribute to excessive vascular calcification. We hypothesize that limiting the accumulation of 7-84 PTH fragments by maintaining a 1-84/7-84 ratio above 1.6 will reduce the amount of vitamin D analogues administered and ultimately reduce the development of coronary calcification. To investigate this hypothesis, we propose to prospectively treat 50 patients with 1, 25 dihydroxyvitamin D2 where doses are determined by maintaining a 1-84/7-84 ration > 1.6 or by maintaining intact PTH levels between 150-350 pg/ml using existing second generation PTH assays.

4.0 Hypothesis & Objectives

4.1 Hypothesis #1: Clinical management of secondary hyperparathyroidism in new hemodialysis patients using the Scantibodies 1-84/7-84 PTH ratio for one year will reduce the amount of Vitamin D administration resulting in reduced coronary calcification compared to patients in which PTH management is accomplished by conventional, second generation PTH assay.

4.1a Specific Aim #1 Specific Aim #1 will compare the amount of coronary calcification and the percentage of patients with at least one coronary lesion > 50% luminal obstruction at baseline and after one-year therapy following randomization to one of two treatment groups.

[Group 1] Patients randomized to group 1 will have the administration of 1alpha OH vitamin D2 (Hectorol) targeted to achieve serum PTH levels between 150-300 ng/ml using a Bayer Centaur iPTH assay.

[Group 2] Patients randomized to group 2 will have the administration of vitamin D analogues targeted to achieve a ratio of 1-84/7-84 PTH fragments between ranges of 1.4-1.6 using the Scantibodies IRMA PTH assay. (Hectorol).

Rationale: Coronary calcification is a frequent complication of end stage renal disease (ESRD) with recent estimates of up to 80% of chronic hemodialysis patients exhibiting moderate to severe vascular calcification 1. Numerous clinical factors have been associated with the development of arterial calcification including hyperphosphatemia 2, diabetes mellitus 3 and calcium containing phosphate binders 4. More recently, the increased use of vitamin D analogues to treat secondary hyperparathyroidism has been implicated as a major contributor to vascular calcification among ESRD patients.

These clinical practices are complicated by the observation that carboxy fragments of PTH (e.g. 7-84) cross react with second generation PTH assays. Because carboxy PTH fragments are either inert or antagonize functional bio-intact PTH (1-84), clinicians have used excessive doses of vitamin D analogues to regulate PTH levels. Moreover, there are animal model studies that suggest that carboxy PTH fragments directly contribute to vascular calcification 16.We propose that clinical decision making using the incomplete information provided the currently available second generation PTH assays leads to excessive vitamin D administration and subsequent acceleration of coronary calcification.

Anticipated Results: We anticipate that prolonged (1 year) management of PTH levels using a second generation of PTH assays will lead to an increase in the total administered dose of vitamin D analogues. Moreover, this increase in vitamin D administration will result in increased coronary calcification at the end of one year of therapy. Conversely, maintaining a 1-84/7-84 PTH ratio between 1.4-1.6 using the Scantibodies third generation assay will reduce the amount of administered vitamin D analogues and subsequently reduce the amount of coronary calcification at one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age > 18 and < 80 years of age
2. Patients receiving outpatient hemodialysis for > 3 or <24 months duration
3. Patients must have baseline coronary calcification defined as at one ROI (regions of interest with >130 Hounsfield units) in 1 or more coronary vessels
4. Patients must have a stable dose of phosphate binder for 30 days prior to study enrollment

Exclusion Criteria:

1. Patients intact PTH < 100 or > 1000 pg/ml
2. Patients on peritoneal dialysis
3. Patients with a previous parathyroidectomy
4. Patients with dry weight > 300 lbs
5. Patients with chronic atrial flutter or fibrillation
6. Patients receiving chronic coumadin therapy
7. Patients with known allergies to contrast dyes
8. Patients receiving current Cinacalcet therapy or during previous 30 days
9. Patients unable to take Metoprolol therapy
10. Patients with resting heart rate >100 and unresponsive to beta blockade
11. Patients with known pregnancy or unwilling to use contraception during the course of the study
12. Patients unable to tolerate the confines of CT scanner
13. Patients with a renal transplant within the previous 5 years
14. Patients with known aluminum toxicity
15. Patients undergoing recent PTCA or CABG within the previous 12 months
16. Patients with ESRD secondary to Sarcoidosis
17. Patients unwilling to use Selevamer as a primary phosphate binder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percent Change in Hounsfield units of coronary calcification between baseline and after one year of therapy | 12 months

SECONDARY OUTCOMES:
Mean dose of Vitamin D2 administered over 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tumlin, MD, Principal Investigator — Southeast Renal Research Institute
Locations (1):
- Davita East Charlotte Dialysis Unit, Charlotte, North Carolina, United States